CLINICAL TRIAL: NCT00969397
Title: Combined Use of Pulsed Dye Laser and Topical Antiangiogenic Agents for Treatment of Port Wine Stain Birthmarks
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: We have decided not to pursue the study
Sponsor: University of California, Irvine (Other)
Collaborators: Beckman Laser Institute University of California Irvine (Other)
Responsible Party: Principal Investigator, Beckman Laser Institute and Medical Center, J S Nelson, M.D., Ph.D.,Professor of Surgery and Biomedical Engineering, University of California, Irvine
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20097069
Record Dates: First submitted 2009-08-31; First posted 2009-09-01 (Estimated); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Port Wine Stain
Keywords: Birthmark; PWS
MeSH Terms: conditions — Port-Wine Stain | interventions — Angiogenesis Inhibitors; Lasers, Dye

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Topical Antiangiogenic (Experimental): Topical Antiangiogenic Agents
  Interventions: Drug: Topical Antiangiogenic
- Pulsed Dye Laser (Experimental): Pulsed Dye Laser
  Interventions: Device: Pulsed Dye Laser

INTERVENTIONS:
Drug: Topical Antiangiogenic — Topical Antiangiogenic
  Arms: Topical Antiangiogenic
Device: Pulsed Dye Laser — Pulsed Dye Laser
  Arms: Pulsed Dye Laser

SUMMARY:
The researcher want to improve port wine stain (PWS) therapeutic outcome in response to laser therapy. The researcher want to determine whether the combined use of pulsed dye laser (PDL) therapy and topical tacrolimus or pimecrolimus will improve PWS therapeutic outcome.

DETAILED DESCRIPTION:
Both topical agents inhibit nuclear factor of activated T-cells (NFAT) which blocks the calcineurin/NFAT pathway inhibiting endothelial cell proliferation and angiogenesis, which could be very useful in preventing PWS recanalization.

The combined use of PDL to induce PWS blood vessel injury, and topical antiangiogenic agents to prevent PWS blood vessel angiogenesis and recanalization after laser therapy, will improve PWS lesion blanching.

ELIGIBILITY:
Inclusion Criteria:

* 16 years of age and older
* Have PWS suitable for comparison testing as determined by the study doctor

Exclusion Criteria:

* Less than 16 years old
* Are pregnant
* Have skin cancer
* Currently taking immunosuppressive or steroids or photosensitizing drugs
* Current participation in any other investigational drug evaluation
* Concurrent use of known photosensitizing drugs

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-11; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Improve PWS lesion blanching. | 8 weeks

SECONDARY OUTCOMES:
To determine whether the combined use of pulsed dye laser (PDL) therapy and topical agent will improve PWS outcome. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: John S Nelson, M.D,PhD, Principal Investigator — Beckman Laser Institute University of California Irvine